CLINICAL TRIAL: NCT01737164
Title: Effect of Age on Glucose and Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nicolas Musi, MD, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC20100133H; 1R01DK089229-01 (NIH)
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Glucose Metabolism Disorders; Lipid Metabolism Disorders; Metabolic Diseases
Keywords: Glucose; Lipid; Metabolism; Non Diabetic; Healthy
MeSH Terms: conditions — Glucose Metabolism Disorders; Lipid Metabolism Disorders; Metabolic Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise - Older Subjects (Experimental): Subjects aged 65 and higher will perform 16 weeks of moderate intensity exercise
  Interventions: Behavioral: Aerobic Exercise
- Aerobic Exercise - Young Subjects (Experimental): Subjects 18-30 years old will perform 16 weeks of moderate intensity exercise
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise

SUMMARY:
Aging is a major risk factor for the development of type 2 diabetes (T2DM). Approximately 50% of subjects aged ≥65 have diabetes or impaired glucose tolerance, a pre-diabetic state. Purpose: In the proposed study, the investigators will test the hypotheses that the decrease in fat oxidation that occurs in muscle from older human subjects is secondary to an age-mediated reduction in AMPK signaling, in vivo, and that upregulating AMPK signaling through exercise training will result in (and correlate with) increased fat oxidation, reduced intramyocellular lipids, and improved insulin action.

DETAILED DESCRIPTION:
Aging is a major risk factor for the development of type 2 diabetes (T2DM). Approximately 50% of subjects aged ≥65 have diabetes or impaired glucose tolerance, a pre-diabetic state. Skeletal muscle is the main site of insulin-stimulated glucose disposal and aging is characterized by muscle insulin resistance. It has been suggested that the insulin resistance of aging results from an age-related accumulation of intramyocellular lipids which impair insulin action. However, the molecular basis for the accumulation of intramyocellular fat and insulin resistance in the elderly remains unknown. AMP-activated protein kinase (AMPK) is an energy-sensing enzyme whose activation results in increased fatty acid oxidation. Purpose: In the proposed study, we will test the hypotheses that the decrease in fat oxidation that occurs in muscle from older human subjects is secondary to an age-mediated reduction in AMPK signaling, in vivo, and that upregulating AMPK signaling through exercise training will result in (and correlate with) increased fat oxidation, reduced intramyocellular lipids, and improved insulin action. Using a primary human muscle cell culture system, also we will test that hypotheses that reduced AMPK signaling in old myotubes leads to lower fat oxidation (in vitro) and that chemical activation of AMPK in old myotubes to the same level as young muscle cells will restore insulin action and help prevent fat-induced insulin resistance. To test these hypotheses the following specific aims (objectives) are proposed:

Specific Aim 1) To determine whether reduced AMPK signaling in muscle from older subjects, in vivo, is associated with lower fat oxidation rates and insulin resistance, and whether physical activity improves glucose homeostasis in older subjects by upregulating AMPK signaling in muscle. We will test the hypotheses that (i) reductions in AMPK signaling in muscle from older subjects will be associated with (predict) lower fat oxidation rates and insulin resistance, in vivo; and (ii) training-induced increases in AMPK signaling in older subjects will be associated with (predict) increases in fat oxidation, reductions in intramyocellular lipids, and improvements in insulin action/sensitivity.

Specific Aim 2) To determine whether age-related declines in AMPK signaling are involved in the reductions in fat oxidation and insulin resistance that occur in aging. Using an in vitro primary muscle cell culture system, we will test the hypotheses that (i) reduced AMPK signaling in myotubes from older subjects leads to decreased mitochondrial fatty acid oxidation; and (ii) reduced AMPK signaling and fat oxidation in myotubes from older subjects will result in increased susceptibility to fat-induced insulin resistance.

Specific Aim 3) To examine whether the age-related reductions in fat oxidation and insulin sensitivity in old muscle cells can be reversed by upregulating AMPK signaling. We will test the hypothesis that chemical activation of AMPK in old myotubes (in vitro) to the same level as young muscle cells will restore insulin signaling and help prevent fat-induced insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. healthy, normally active, younger (18-30 y), normal glucose tolerant subjects, without a family history of T2DM (neither parent nor siblings), and BMI of 23-26 kg/m2.
2. healthy, normally active, older (≥65 y), normal glucose tolerant subjects without a family history of T2DM, and BMI of 23-26 kg/m2.
3. Women must be non-lactating. Female patients are eligible only if they have a negative pregnancy test throughout the study period (or postmenopausal). Postmenopausal women taking hormone replacement will be included if they have been on a stable dose for ≥6 months. In younger menstruating woman, all metabolic studies will be performed on the follicular phase of the menstrual cycle.
4. Subjects must have the following laboratory values: Hematocrit ≥ 35%, serum creatinine ≤ 1.5 mg/dl, AST < 2 X upper limit of normal, ALT < 2 X upper limit of normal, alkaline phosphatase < 2 X upper limit of normal, normal urinalysis, and normal platelets, PT and PTT.

Exclusion Criteria:

1. Subjects with diabetes or impaired glucose tolerance based on ADA criteria.
2. Subjects taking drugs known to affect glucose and lipid homeostasis will be excluded.
3. Patients with a history of heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the ECG), peripheral vascular disease, or pulmonary disease.
4. Recent pulmonary embolus, poorly controlled blood pressure (systolic BP>170, diastolic BP>95), resting heart rate >100, electrolyte abnormalities, neuromuscular or musculoskeletal disease.
5. Subjects who smoke.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-09; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Effect of Age on Glucose and Lipid Metabolism | 16 weeks
  Effect of Age on Glucose and Lipid Metabolism; Measurement of glucose and lipid metabolism will be done pre and post exercise in two groups (younger and older subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Musi, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Texas Diabetes Insitute, San Antonio, Texas, United States